CLINICAL TRIAL: NCT03977974
Title: A Safety, Tolerability, Pharmacokinetic, and Pilot Food Effect Study of Single- and Multiple-Ascending Doses of LY3526318 in Healthy Participants
Brief Title: A Study of LY3526318 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID-19 pandemic.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17426; J2D-MC-CVAA (Other: Eli Lilly and Company); 2019-001902-80 (EudraCT Number)
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LY3526318 - Part A (Experimental): Single-ascending dose (SAD) 10 milligram (mg), 30 mg, 50 mg, or 300 mg LY3526318 administered orally.
  100 mg LY3526318 administered orally without a meal in period 1 and 30 mg LY3526318 administered orally with a meal in period 2.
  200 mg LY3526318 administered orally without a meal in period 1 and 200 mg LY3526318 administered orally with a meal in period 2.
  100 mg LY3526318 Fed:
  Period 1: 100 mg LY3526318 administered orally 30 minutes (min) after breakfast (Fed (-30 min.)).
  Period 2: 100 mg LY3526318 orally 30 minutes before breakfast (Fed (+30 min.)).
  Period 3: 100 mg LY3526318 administered orally 60 minutes before breakfast (Fed (+60 min.)).
  Placebo Fed:
  Period 1: Placebo administered orally 30 minutes after breakfast (Fed (-30 min.)).
  Period 2: Placebo administered orally 30 minutes before breakfast (Fed (+30 min.)).
  Period 3: Placebo administered orally 60 minutes before breakfast (Fed (+60 min.)).
  Interventions: Drug: LY3526318
- Placebo - Part A (Placebo Comparator): Participants received placebo administered orally once.
  Interventions: Drug: Placebo
- LY3526318 - Part B (Experimental): Multiple-ascending dose (MAD): 30 mg LY3526318 once daily (QD):
  Participants received 30 mg LY3526318 QD administered orally for 14 days.
  MAD: 60 mg LY3526318 QD:
  Participants received 60 mg LY3526318 QD administered orally for 14 days.
  MAD: 100 mg LY352631 QD:
  Participants received 100 mg LY3526318 QD administered orally for 14 days.
  Interventions: Drug: LY3526318
- Placebo - Part B (Placebo Comparator): Participants received placebo QD orally for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3526318 — Administered orally
  Arms: LY3526318 - Part A; LY3526318 - Part B
Drug: Placebo — Administered orally
  Arms: Placebo - Part A; Placebo - Part B

SUMMARY:
The main purpose of this study is to learn more about the safety and side effects of LY3526318 when given by mouth to healthy participants. The study will have two parts. Each participant will enroll in only one part. For each participant, Part A will last up to 28 days and Part B will last up to 51 days, including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Part A Cohorts:

- Healthy male participants (including self-reported surgically sterile males) must agree to the following:

* When engaging in sex with Women of Child-Bearing Potential (WOCBP) both the male participant and his female partner must use highly effective contraception consisting of 2 forms of birth control (1 of which must be a male barrier method such as a latex or polyurethane condom) from start of dosing throughout the clinical study period, and for 90 days after the final study drug administration
* Nonsurgically sterile male participants must not donate sperm at any time from start of dosing until 90 days beyond the administration of study drug

All Part A and Part B Cohorts:

* Female participants must be nonpregnant and not lactating, or of nonchildbearing potential (either surgically sterilized [e.g. tubal occlusion, hysterectomy, bilateral salpingectomy] or physiologically incapable of becoming pregnant, or postmenopausal with amenorrhea for at least 12 consecutive months). Healthy female participants of child-bearing potential who have a fertile male sexual partner must be willing and able to practice effective contraception from admission to 30 days after the final visit. Sexually active participants must use a combination of 2 of the following methods of contraception, including at least 1 so-called 'barrier' method:

  * Hormonal contraceptive (oral, transdermal patches, vaginal or injectable)
  * Intrauterine device with or without hormones
  * Condom ('barrier' method)
  * Diaphragm or cervical cap
  * Sexual abstinence
* Have a body mass index 18 to 32 kilograms per square meter (kg/m²)

Exclusion Criteria:

* Are currently enrolled in a clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have a history or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, convulsions, or any clinically significant laboratory abnormality
* In the opinion of the investigator are considered to be a danger to themselves
* Have an abnormality in the 12-lead electrocardiogram (ECG)
* Have a history of clinically significant multiple or severe drug allergies or severe post treatment hypersensitivity reactions
* Have donated blood of more than 500 milliliter (mL) within the previous month
* Are unwilling to stop alcohol and caffeinated beverage consumption and smoking/use of tobacco while resident in the CRU
* Have an average weekly alcohol intake that exceeds 21 units per week (1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits
* Have an abnormal blood pressure
* Participants with a history of drug abuse
* Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer)
* Are unwilling to comply with the required dietary restrictions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consists of 2 parts:
  * Part A: Single-ascending dose (SAD, [including a food effect (FE)]).
  * Part B: Multiple-ascending dose (MAD).
  Both parts were randomized, double-blind, and placebo-controlled, with the exception of the 100 milligram (mg) FE part.
Groups:
- SAD: Placebo: Participants received placebo administered orally.
- SAD: 10 mg LY3526318: Participants received 10 mg LY3526318 administered orally.
- SAD: 30 mg LY3526318: Participants received 30 mg LY3526318 administered orally.
- SAD: 50 mg LY3526318: Participants received 50 mg LY3526318 administered orally.
- SAD: 100 mg LY3526318 (Fasted) and 30 mg LY3526318 (Fed): Period 1:
  Participants received 100 mg LY3526318 administered orally without a meal.
  Period 2:
  Participants received 30 mg LY3526318 administered orally with a meal.
- SAD: 200 mg LY3526318 (Fasted) and 200 mg LY3526318 (Fed): Period 1:
  Participants received 200 mg LY3526318 administered orally without a meal.
  Period 2:
  Participants received 200 mg LY3526318 administered orally with a meal.
- SAD: 300 mg LY3526318: Participants received 300 mg LY3526318 administered orally.
- SAD: 100 mg LY3526318 Fed: Period 1: Participants received 100 mg LY3526318 administered orally 30 minutes after breakfast (Fed [-30 min.])
  Period 2:
  Participants received 100 mg LY3526318 orally 30 minutes before breakfast (Fed [+30 min.])
  Period 3: Participants received 100 mg LY3526318 administered orally 60 minutes before breakfast (Fed [+60 min.])
- SAD: Placebo Fed: Period 1: Participants received placebo administered orally 30 minutes after breakfast (Fed [-30 min.])
  Period 2:
  Participants received placebo administered orally 30 minutes before breakfast (Fed [+30 min.])
  Period 3: Participants received placebo administered orally 60 minutes before breakfast (Fed [+60 min.])
- MAD: Placebo QD: Participants received placebo once daily (QD) administered orally for 14 days.
- MAD: 30 mg LY3526318 QD: Participants received 30 mg LY3526318 QD administered orally for 14 days.
- MAD: 60 mg LY3526318 QD: Participants received 60 mg LY3526318 QD administered orally for 14 days.
- MAD: 100 mg LY352631 QD: Participants received 100 mg LY3526318 QD administered orally for 14 days.
Period: Period 1
Arm/Group | SAD: Placebo | SAD: 10 mg LY3526318 | SAD: 30 mg LY3526318 | SAD: 50 mg LY3526318 | SAD: 100 mg LY3526318 (Fasted) and 30 mg LY3526318 (Fed) | SAD: 200 mg LY3526318 (Fasted) and 200 mg LY3526318 (Fed) | SAD: 300 mg LY3526318 | SAD: 100 mg LY3526318 Fed | SAD: Placebo Fed | MAD: Placebo QD | MAD: 30 mg LY3526318 QD | MAD: 60 mg LY3526318 QD | MAD: 100 mg LY352631 QD
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 1 | 6 | 6 | 6 | 6
Received at Least One Dose of Study Drug | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 1 | 6 | 6 | 6 | 6
Completed | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 1 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | SAD: Placebo | SAD: 10 mg LY3526318 | SAD: 30 mg LY3526318 | SAD: 50 mg LY3526318 | SAD: 100 mg LY3526318 (Fasted) and 30 mg LY3526318 (Fed) | SAD: 200 mg LY3526318 (Fasted) and 200 mg LY3526318 (Fed) | SAD: 300 mg LY3526318 | SAD: 100 mg LY3526318 Fed | SAD: Placebo Fed | MAD: Placebo QD | MAD: 30 mg LY3526318 QD | MAD: 60 mg LY3526318 QD | MAD: 100 mg LY352631 QD
Started | 0 (Period 2 does not apply to this arm.) | 0 (Period 2 does not apply to this arm.) | 0 (Period 2 does not apply to this arm.) | 0 (Period 2 does not apply to this arm.) | 6 | 6 | 0 (Period 2 does not apply to this arm.) | 3 | 1 | 0 (Period 2 does not apply to this arm.) | 0 (Period 2 does not apply to this arm.) | 0 (Period 2 does not apply to this arm.) | 0 (Period 2 does not apply to this arm.)
Completed | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | SAD: Placebo | SAD: 10 mg LY3526318 | SAD: 30 mg LY3526318 | SAD: 50 mg LY3526318 | SAD: 100 mg LY3526318 (Fasted) and 30 mg LY3526318 (Fed) | SAD: 200 mg LY3526318 (Fasted) and 200 mg LY3526318 (Fed) | SAD: 300 mg LY3526318 | SAD: 100 mg LY3526318 Fed | SAD: Placebo Fed | MAD: Placebo QD | MAD: 30 mg LY3526318 QD | MAD: 60 mg LY3526318 QD | MAD: 100 mg LY352631 QD
Started | 0 (Period 3 does not apply to this arm.) | 0 (Period 3 does not apply to this arm.) | 0 (Period 3 does not apply to this arm.) | 0 (Period 3 does not apply to this arm.) | 0 (Period 3 does not apply to this arm.) | 0 (Period 3 does not apply to this arm.) | 0 (Period 3 does not apply to this arm.) | 3 | 1 | 0 (Period 3 does not apply to this arm.) | 0 (Period 3 does not apply to this arm.) | 0 (Period 3 does not apply to this arm.) | 0 (Period 3 does not apply to this arm.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- MAD: Placebo QD: Participants received placebo one daily (QD) administered orally for 14 days.
- Total: Total of all reporting groups
Arm/Group | SAD: Placebo | SAD: 10 mg LY3526318 | SAD: 30 mg LY3526318 | SAD: 50 mg LY3526318 | SAD: 100 mg LY3526318 (Fasted) and 30 mg LY3526318 (Fed) | SAD: 200 mg LY3526318 (Fasted) and 200 mg LY3526318 (Fed) | SAD: 300 mg LY3526318 | SAD: 100 mg LY3526318 Fed | SAD: Placebo Fed | MAD: Placebo QD | MAD: 30 mg LY3526318 QD | MAD: 60 mg LY3526318 QD | MAD: 100 mg LY352631 QD | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 1 | 6 | 6 | 6 | 6 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (17) | 41 (20) | 30 (17) | 26 (3) | 36 (20) | 39 (14) | 40 (19) | 46 (21) | 49 (NA) — There is no SD for N=1. | 35 (8) | 38 (14) | 29 (14) | 35 (15) | 35.09 (15.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 6 | 3 | 6 | 6 | 6 | 3 | 1 | 6 | 6 | 6 | 6 | 70
  Male | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 6
  Not Hispanic or Latino | 12 | 6 | 5 | 5 | 4 | 6 | 6 | 3 | 1 | 6 | 5 | 6 | 5 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 5
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 10 | 6 | 5 | 5 | 5 | 5 | 5 | 2 | 1 | 3 | 4 | 5 | 4 | 60
  More than one race | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 1 | 6 | 6 | 6 | 6 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is any AE from this study that results in 1 of the following: death, initial or prolonged inpatient hospitalization, a life-threatening experience (i.e. immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly/birth defect and important medical events that may not be immediately life threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent 1 of the other outcomes listed in the definition. A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, are reported in the Adverse Events module section.
Time Frame: Baseline Up To 32 Days
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- SAD: 50 mg LY3526318: Participants received 50 mg LY3526318 orally.
- MAD: Placebo QD: Participants received placebo one daily (QD) orally for 14 days.
Arm/Group | SAD: Placebo | SAD: 10 mg LY3526318 | SAD: 30 mg LY3526318 | SAD: 50 mg LY3526318 | SAD: 100 mg LY3526318 (Fasted) and 30 mg LY3526318 (Fed) | SAD: 200 mg LY3526318 (Fasted) and 200 mg LY3526318 (Fed) | SAD: 300 mg LY3526318 | SAD: 100 mg LY3526318 Fed | SAD: Placebo Fed | MAD: Placebo QD | MAD: 30 mg LY3526318 QD | MAD: 60 mg LY3526318 QD | MAD: 100 mg LY352631 QD
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 1 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3526318
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3526318
Time Frame: SAD: Day 1: predose, 1, 2, 4, 6, 8 and 12 hours postdose; Day 2 and Day 3: 24 and 48 hours postdose; 3-Period Food Effect Arms: Day 1: Predose, 1, 2, 4, 6, 8 and 12 hours, Day 2, Day 3 and Day 4: Predose, 24, 48 and 72 hours postdose
Population: SAD: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- SAD: 100 mg LY3526318: Participants received 100 mg LY3526318 administered orally without a meal.
- SAD: 200 mg LY3526318: Participants received 200 mg LY3526318 administered orally without a meal.
- SAD: 30 mg LY3526318 Fed: Participants received 30 mg LY3526318 administered orally with a meal.
- SAD: 200 mg LY3526318 Fed: Participants received 200 mg LY3526318 administered orally with a meal.
- SAD FE : 100 mg LY3526318 Fed (-30 Min): Participants received 100 mg LY3526318 administered orally 30 minutes after breakfast (Fed [-30 min.]).
- SAD FE: 100 mg LY Fed (+30 Min): Participants received 100 mg LY3526318 orally 30 minutes before breakfast (Fed [+30 min.]).
- SAD FE: 100 mg LY Fed (+60 Min): Participants received placebo administered orally 60 minutes before breakfast (Fed [+60 min.])
Arm/Group | SAD: 10 mg LY3526318 | SAD: 30 mg LY3526318 | SAD: 50 mg LY3526318 | SAD: 100 mg LY3526318 | SAD: 200 mg LY3526318 | SAD: 300 mg LY3526318 | SAD: 30 mg LY3526318 Fed | SAD: 200 mg LY3526318 Fed | SAD FE : 100 mg LY3526318 Fed (-30 Min) | SAD FE: 100 mg LY Fed (+30 Min) | SAD FE: 100 mg LY Fed (+60 Min)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 4 | 6 | 1 | 4 | 2 | 3 | 3
nanogram*hour per milliliter (ng*h/mL) | 2322 (64.3) | 6132 (107.0) | 15442 (63.6) | 55533 (56.6) | 45746 (58.5) | 58311 (100.3) | NA (NA) — Geometric mean and coefficient of variation couldn't be calculated as there was only a single participant. Individual value reported = 7058 ng*h/mL. | 10603 (107.0) | 6379 (47.4) | 19028 (15.3) | 20237 (38.8)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to 24 Hours (AUC[0-24]) of LY3526318
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to 24 hours (AUC[0-24]) of LY3526318
Time Frame: MAD: Day 1: Predose,1, 2, 4, 6, 8 and 12 hours post dose
Population: MAD: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MAD: 30 mg LY3526318 QD | MAD: 60 mg LY3526318 QD | MAD: 100 mg LY352631 QD
Number analyzed (Participants) | 6 | 6 | 6
ng*h/mL | 6015 (80.7) | 18525 (48.1) | 25769 (68.4)

4. Secondary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of LY3526318
Description: PK: Maximum Observed Drug Concentration (Cmax) of LY3526318
Time Frame: as for outcome 2
Population: SAD: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | SAD: 10 mg LY3526318 | SAD: 30 mg LY3526318 | SAD: 50 mg LY3526318 | SAD: 100 mg LY3526318 | SAD: 200 mg LY3526318 | SAD: 300 mg LY3526318 | SAD: 30 mg LY3526318 Fed | SAD: 200 mg LY3526318 Fed | SAD FE : 100 mg LY3526318 Fed (-30 Min) | SAD FE: 100 mg LY Fed (+30 Min) | SAD FE: 100 mg LY Fed (+60 Min)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 3 | 3 | 3
nanogram per milliliter (ng/mL) | 188 (100.7) | 573 (119.5) | 1321 (58.9) | 4265 (60.8) | 5047 (40.6) | 4879 (120.8) | 204 (51.6) | 719 (139.0) | 378 (43.3) | 1288 (34.9) | 1407 (91.2)

5. Secondary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of LY3526318
Description: PK: Maximum Observed Drug Concentration (Cmax) of LY3526318
Time Frame: MAD: Day 1 and Day 14: Predose, 1, 2, 4, 6, 8 and 12 hours post dose
Population: MAD: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MAD: 30 mg LY3526318 QD | MAD: 60 mg LY3526318 QD | MAD: 100 mg LY352631 QD
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Day 1 | 666 (92.5) | 2117 (35.7) | 2987 (60.6)
  Day 14 | 1017 (39.7) | 2791 (63.2) | 4224 (38.1)

6. Secondary Outcome: PK: Time to Maximum Concentration (Tmax) of LY3526318
Description: PK: Time to Maximum Concentration (Tmax) of LY3526318
Time Frame: as for outcome 2
Population: SAD: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | SAD: 10 mg LY3526318 | SAD: 30 mg LY3526318 | SAD: 50 mg LY3526318 | SAD: 100 mg LY3526318 | SAD: 200 mg LY3526318 | SAD: 300 mg LY3526318 | SAD: 30 mg LY3526318 Fed | SAD: 200 mg LY3526318 Fed | SAD FE : 100 mg LY3526318 Fed (-30 Min) | SAD FE: 100 mg LY Fed (+30 Min) | SAD FE: 100 mg LY Fed (+60 Min)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 3 | 3 | 3
hours | 2.03 [2.00 to 4.02] | 2.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 4.00 [2.00 to 4.02] | 4.00 [2.00 to 4.02] | 4.00 [2.00 to 4.00] | 12.00 [4.00 to 24.02] | 4.00 [2.00 to 8.02] | 4.03 [4.03 to 12.00] | 4.00 [1.00 to 4.08] | 4.00 [2.00 to 12.00]

7. Secondary Outcome: PK: Time to Maximum Concentration (Tmax) of LY3526318
Description: PK: Time to Maximum Concentration (Tmax) of LY3526318
Time Frame: MAD: Day 1 and Day 14: Predose, 1, 2, 4, 6, 8 and 12 hours post dose
Population: MAD: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | MAD: 30 mg LY3526318 QD | MAD: 60 mg LY3526318 QD | MAD: 100 mg LY352631 QD
Number analyzed (Participants) | 6 | 6 | 6
hours
  Day 1 | 4.00 [2.00 to 24.00] | 3.00 [2.00 to 4.02] | 3.00 [2.00 to 4.03]
  Day 14 | 4.01 [2.00 to 4.03] | 4.01 [2.00 to 4.03] | 4.00 [2.00 to 4.03]

ADVERSE EVENTS:
Time Frame: Baseline Up To 32 Days
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- SAD: 100 mg LY Fed (-30 Min): Participants received 100 mg LY3526318 administered orally 30 minutes after breakfast (Fed [-30 min.])
- SAD: 100 mg LY Fed (+30 Min): Participants received 100 mg LY3526318 orally 30 minutes before breakfast (Fed [+30 min.])
- SAD:100 mg LY Fed (+60 Min): Participants received 100 mg LY3526318 administered orally 60 minutes before breakfast (Fed [+60 min.]).
- SAD: Placebo Fed (-30 Min): Participants received placebo administered orally 30 minutes after breakfast (Fed [-30 min.]).
- SAD: Placebo Fed (+30 Min): Participants received placebo administered orally 30 minutes before breakfast (Fed [+30 min.]).
- SAD: Placebo Fed (+60 Min): Participants received placebo administered orally 60 minutes before breakfast (Fed [+60 min.]).
- MAD: 30 mg LY3526318 QD LY3526318 QD: Participants received 30 mg LY3526318 QD administered orally for 14 days.
- MAD: 60 mg LY3526318 QD LY3526318 QD: Participants received 60 mg LY3526318 QD administered orally for 14 days.
Arm/Group | SAD: Placebo | SAD: 10 mg LY3526318 | SAD: 30 mg LY3526318 | SAD: 50 mg LY3526318 | SAD: 100 mg LY3526318 | SAD: 200 mg LY3526318 | SAD: 300 mg LY3526318 | SAD: Placebo Fed | SAD: 30 mg LY3526318 Fed | SAD: 200 mg LY3526318 Fed | SAD: 100 mg LY Fed (-30 Min) | SAD: 100 mg LY Fed (+30 Min) | SAD:100 mg LY Fed (+60 Min) | SAD: Placebo Fed (-30 Min) | SAD: Placebo Fed (+30 Min) | SAD: Placebo Fed (+60 Min) | MAD: Placebo QD | MAD: 30 mg LY3526318 QD LY3526318 QD | MAD: 60 mg LY3526318 QD LY3526318 QD | MAD: 100 mg LY352631 QD
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6 | 0/3 | 0/3 | 0/3 | 0/1 | 0/1 | 0/1 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6 | 0/3 | 0/3 | 0/3 | 0/1 | 0/1 | 0/1 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/12 | 2/6 | 5/6 | 0/6 | 4/6 | 2/6 | 3/6 | 1/4 | 2/6 | 0/6 | 3/3 | 3/3 | 1/3 | 1/1 | 1/1 | 1/1 | 6/6 | 5/6 | 4/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | SAD: Placebo (N=12) | SAD: 10 mg LY3526318 (N=6) | SAD: 30 mg LY3526318 (N=6) | SAD: 50 mg LY3526318 (N=6) | SAD: 100 mg LY3526318 (N=6) | SAD: 200 mg LY3526318 (N=6) | SAD: 300 mg LY3526318 (N=6) | SAD: Placebo Fed (N=4) | SAD: 30 mg LY3526318 Fed (N=6) | SAD: 200 mg LY3526318 Fed (N=6) | SAD: 100 mg LY Fed (-30 Min) (N=3) | SAD: 100 mg LY Fed (+30 Min) (N=3) | SAD:100 mg LY Fed (+60 Min) (N=3) | SAD: Placebo Fed (-30 Min) (N=1) | SAD: Placebo Fed (+30 Min) (N=1) | SAD: Placebo Fed (+60 Min) (N=1) | MAD: Placebo QD (N=6) | MAD: 30 mg LY3526318 QD LY3526318 QD (N=6) | MAD: 60 mg LY3526318 QD LY3526318 QD (N=6) | MAD: 100 mg LY352631 QD (N=6)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug withdrawal headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (4) | 2 (2) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomenorrhoea (Reproductive system and breast disorders) | 0/11 (0) | 0/4 (0) | 0 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstrual discomfort (Reproductive system and breast disorders) | 0/11 (0) | 0/4 (0) | 0 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated due to COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT03977974/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT03977974/SAP_001.pdf